CLINICAL TRIAL: NCT03536117
Title: Phase 2a Dose-Defining Safety and Immunogenicity Study of MTBVAC in South African Neonates Living in a High-Burden Tuberculosis-Endemic Region
Brief Title: Dose-Defining Safety and Immunogenicity Study of MTBVAC in South African Neonates
Acronym: MTBVAC-03
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biofabri, S.L (Industry)
Collaborators: South African Tuberculosis Vaccine Initiative (Other); Universidad de Zaragoza (Other); TuBerculosis Vaccine Initiative (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MTBVAC-03
Record Dates: First submitted 2018-02-16; First posted 2018-05-24 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — MTBVAC vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MTBVAC Group 1 (Experimental): MTBVAC intermediate dose 2.5 x 10E+04 CFU/0.05 mL
  Interventions: Biological: MTBVAC
- MTBVAC Group 2 (Experimental): MTBVAC high dose 2.5 x 10E+05 CFU/0.05 mL
  Interventions: Biological: MTBVAC
- MTBVAC Group 3 (Experimental): MTBVAC highest dose 2.5 x 10E+06 CFU/0.05 mL
  Interventions: Biological: MTBVAC
- BCG Group 4 (Active Comparator): BCG control 2.5 x 10E+05 CFU/0.05 mL
  Interventions: Biological: BCG

INTERVENTIONS:
Biological: MTBVAC — Live-attenuated Mycobacterium tuberculosis based on the deletion of phoP and fadD26 virulence genes
  Arms: MTBVAC Group 1; MTBVAC Group 2; MTBVAC Group 3
Biological: BCG — Live-attenuated Mycobacterium bovis obtained by subculture passaging in ox-bile and glycerated potatoes between 1908-1921 by Albert Calmette and Camille Guerin. BCG is the only licensed vaccine today against tuberculosis (TB) mainly used in TB-endemic countries.
  Other Names: Licensed BCG
  Arms: BCG Group 4

SUMMARY:
A Phase 2a dose-defining study of MTBVAC to evaluate the safety, reactogenicity, immunogenicity, and potential for IGRA conversion and reversion, of MTBVAC in South African newborns. Ninety-nine HIV unexposed, BCG naïve newborns will be randomized to receive either BCG 2.5 x 105 CFU (n=24) or MTBVAC at one of three dose levels (n=75). Allocation will be double blind. Enrolment will be sequential into 3 cohorts of increasing MTBVAC dose (Cohort 1: n=25 MTBVAC 2.5 x 10E+04 and n=8 BCG; Cohort 2: n=25 MTBVAC 2.5 x 10E+05 and n=8 BCG; Cohort 3: n=25 MTBVAC 2.5 x 10E+06 and n=8 BCG). Dose escalation will be staggered to allow gradual evaluation of safety; final selection of the dose for Cohort 3 will be based on all available safety and immunogenicity data.

DETAILED DESCRIPTION:
new effective tuberculosis (TB) vaccine is essential to achieve World Health Organization (WHO) End TB goals and eliminate TB by 2050. The optimal long-term strategy would be a combination of serial mass campaigns in adults, coupled with universal newborn vaccination. Newborns are the only human population without prior mycobacterial exposure in TB endemic countries and as such, live attenuated mycobacterial vaccines may offer better protection to this naïve population compared to adults.

MTBVAC is a novel TB vaccine candidate generated by genetically attenuating an M. tuberculosis clinical isolate of the EuroAmerican lineage. MTBVAC is based on two independent, stable genetic deletions of the genes coding for two major virulence factors, phoP coding for the transcription factor PhoP and fadD26 coding for the synthesis of PDIM. Since MTBVAC contains most of the genes deleted from BCG, it presents a wider collection of mycobacterial antigens to the host immune system. Safety and immunogenicity of MTBVAC has been demonstrated in BCG naive adults; and MTBVAC appears safe in a small ongoing Phase 1b study in South African newborns. Definitive demonstration of safety and immunogenicity at the optimal MTBVAC dose is key to progression into multi-centre efficacy trials in newborns.

A Phase 2a dose-defining study of MTBVAC to evaluate the safety, reactogenicity, immunogenicity, and potential for IGRA conversion and reversion, of MTBVAC in South African newborns. Ninety-nine HIV unexposed, BCG naïve newborns will be randomized to receive either BCG 2.5 x 105 CFU (n=24) or MTBVAC at one of three dose levels (n=75). Allocation will be double blind. Enrolment will be sequential into 3 cohorts of increasing MTBVAC dose (Cohort 1: n=25 MTBVAC 2.5 x 10E+04 and n=8 BCG; Cohort 2: n=25 MTBVAC 2.5 x 10E+05 and n=8 BCG; Cohort 3: n=25 MTBVAC 2.5 x 10E+06 and n=8 BCG). Dose escalation will be staggered to allow gradual evaluation of safety; final selection of the dose for Cohort 3 will be based on all available safety and immunogenicity data.

ELIGIBILITY:
Inclusion Criteria of Newborns:

* Newborns of mothers who provided informed consent will be enrolled within 96 hours of birth if they are in general good health during pregnancy and delivery
* Weight ≥2450 grams at birth
* Apgar score at 5 minutes ≥7
* Estimated gestational age ≥37 weeks.

Exclusion Criteria of Newborns:

* If received routine BCG vaccination prior to enrolment
* Have any significant antenatal or intrapartum or postpartum complications
* Have unknown or positive maternal HIV test; or
* Have prior history of close contact with a TB patient, antenatal or postnatal, whether maternal, other family member or other household member.

Max Age: 96 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 99 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2022-05-17 (Actual); Study Completion 2022-05-17 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as defined in protocol. | 365 days post-vaccination
  * Solicited systemic adverse events: fever, irritability, vomiting, diarrhea, drowsiness, poor feeding, skin rash.
  * Solicited injection site reaction adverse events: pain, redness, swelling, ulceration, drainage, and regional lymphadenopathy
  * Unsolicited adverse events and serious adverse events
Immunogenicity analysis in infants | 365 days post-vaccination
  Measure of CD4 and CD8 T cells expressing specific cytokines in whole blood.

SECONDARY OUTCOMES:
MTBVAC-induced QFT conversion and reversion kinetics | 365 days post-vaccination
  Quantitative and qualitative results of the QFT Gold Plus assay up to day 365 post-vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Tameris, MD, Principal Investigator — Study Principal Investigator South African Tuberculosis Vaccine Initiative
Locations (1):
- SATVI: Worcester, Worcester, Western Cape, South Africa

REFERENCES:
- [Background] Arbues A, Aguilo JI, Gonzalo-Asensio J, Marinova D, Uranga S, Puentes E, Fernandez C, Parra A, Cardona PJ, Vilaplana C, Ausina V, Williams A, Clark S, Malaga W, Guilhot C, Gicquel B, Martin C. Construction, characterization and preclinical evaluation of MTBVAC, the first live-attenuated M. tuberculosis-based vaccine to enter clinical trials. Vaccine. 2013 Oct 1;31(42):4867-73. doi: 10.1016/j.vaccine.2013.07.051. Epub 2013 Aug 17. PMID 23965219
- [Background] Spertini F, Audran R, Chakour R, Karoui O, Steiner-Monard V, Thierry AC, Mayor CE, Rettby N, Jaton K, Vallotton L, Lazor-Blanchet C, Doce J, Puentes E, Marinova D, Aguilo N, Martin C. Safety of human immunisation with a live-attenuated Mycobacterium tuberculosis vaccine: a randomised, double-blind, controlled phase I trial. Lancet Respir Med. 2015 Dec;3(12):953-62. doi: 10.1016/S2213-2600(15)00435-X. Epub 2015 Nov 17. PMID 26598141
- [Background] Aguilo N, Uranga S, Marinova D, Monzon M, Badiola J, Martin C. MTBVAC vaccine is safe, immunogenic and confers protective efficacy against Mycobacterium tuberculosis in newborn mice. Tuberculosis (Edinb). 2016 Jan;96:71-4. doi: 10.1016/j.tube.2015.10.010. Epub 2015 Nov 30. PMID 26786657
- [Background] Clark S, Lanni F, Marinova D, Rayner E, Martin C, Williams A. Revaccination of Guinea Pigs With the Live Attenuated Mycobacterium tuberculosis Vaccine MTBVAC Improves BCG's Protection Against Tuberculosis. J Infect Dis. 2017 Sep 1;216(5):525-533. doi: 10.1093/infdis/jix030. PMID 28329234
- [Background] Marinova D, Gonzalo-Asensio J, Aguilo N, Martin C. MTBVAC from discovery to clinical trials in tuberculosis-endemic countries. Expert Rev Vaccines. 2017 Jun;16(6):565-576. doi: 10.1080/14760584.2017.1324303. Epub 2017 May 12. PMID 28447476
- [Result] Tameris M, Rozot V, Imbratta C, Geldenhuys H, Mendelsohn SC, Kany Luabeya AK, Shenje J, Tredoux N, Fisher M, Mulenga H, Bilek N, Young C, Veldsman A, Botes N, Thole J, Fritzell B, Mukherjee R, Jelsbak IM, Rodriguez E, Puentes E, Doce J, Marinova D, Gonzalo-Asensio J, Aguilo N, Martin C, Scriba TJ, Hatherill M; MTBVAC 202 study team. Safety, reactogenicity, and immunogenicity of MTBVAC in infants: a phase 2a randomised, double-blind, dose-defining trial in a TB endemic setting. EBioMedicine. 2025 Apr;114:105628. doi: 10.1016/j.ebiom.2025.105628. Epub 2025 Mar 17. PMID 40101388

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-15): https://cdn.clinicaltrials.gov/large-docs/17/NCT03536117/Prot_SAP_000.pdf